CLINICAL TRIAL: NCT02715310
Title: Haemodynamic Monitoring in Head and Neck Cancer Patients
Acronym: HMHN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: MKG HN 1
Record Dates: First submitted 2016-03-07; First posted 2016-03-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood parameters
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to estimate the effect of fluid management in regard to postoperative complications this observatory study will document every kind of fluid intervention peri- and intraoperatively.

DETAILED DESCRIPTION:
The extend of mass transfusions is known to correlate with postoperative complications. However, also crystalloid and colloidal infusions are under suspicion to cause postoperative complications. This study will capture any kind of fluid intervention perioperatively as well as intraoperatively. Intraoperative fluid management will be documented and matched with the operation steps respectively. The extend of fluid therapy will be correlated with general postoperative complications and especially with the survival of microvascular transplants.

For this purpose, there will be four questionaires. After informed consent, the first questionaire will cover the patient's history, risk factors and previous operations. The second questionaire will cover intraoperative fluid management, documented with the actual operation step. Furthermore, it will also intraoperative complications, cardiovascular-active medication. For closer monitoring, data from Picco will also be included. The third questionaire will be complete in the ICU covering similar content as the second questionaire. The last questionaire will cover the patient's progress on the general ward. Fluid management and tube feeding, as well as general postoperative complication and flap specific complications will be noted.

This study aims for 50-80 patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* admitted for head and neck surgery with microvascular transplantation due to head and neck tumors

Exclusion Criteria:

* Pregnancy
* underage
* missing informed consent
* revisions and relapse operations
* non tumor-associated operations
* surgery without microvascular transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Full grown, able to consent patients admitted for major head and neck surgery with planned microvascular transplants for reconstruction due to tumors in the head and neck region.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 1 week
  General Complications e.g. affecting lung, cardiovascular system, kidneys

SECONDARY OUTCOMES:
Transplant Survival via Clinical Examination | One week
  Transplant Survival via Clinical Examination/ Need for further microvascular Transplant

CONTACTS AND LOCATIONS:
Overall Officials: Denys Loeffelbein, PhD, MD, DDS, Study Chair — Technical University Muncih
Locations (1):
- Department of Oral and Maxillofacial Surgery, Technische Universität München, Munich, Bavaria, Germany